CLINICAL TRIAL: NCT07214688
Title: A Phase 2 Study of Fludarabine and Intermediate-dose Total Body Irradiation (800 cGy) Followed by Post-transplant Cyclophosphamide in Patients Aged 18-65 Undergoing Allogeneic Stem Cell Transplant for Hematologic Malignancies
Brief Title: Fludarabine and Intermediate-dose TBI Followed by PTCy in Patients Undergoing Allo Transplant for Heme Malignancies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLU-TBI-800-PTCY; Pro2025-0254 (Other: HMH)
Record Dates: First submitted 2025-10-03; First posted 2025-10-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Allogeneic Stem Cell Transplant Recipient
MeSH Terms: interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental (Experimental): Fludarabine and Intermediate-dose Total Body Irradiation (800 cGy) Followed by Post-transplant Cyclophosphamide
  Interventions: Drug: Fludarabine; Radiation: Intermediate-dose Total Body Irradiation (TBI); Drug: Post-transplant Cyclophosphamide (PTCy); Drug: Tacrolimus; Drug: Mycophenolate mofetil (MMF)

INTERVENTIONS:
Drug: Fludarabine — Patients will receive fludarabine administered at the dose of 30 mg/m2 intravenously daily on Days -6 to -2
  Other Names: Fludara; Oforta
Radiation: Intermediate-dose Total Body Irradiation (TBI) — Patients will receive intermediate-dose total body irradiation (TBI) administered at the dose of 800 cGy in 4 total fractions, 2 fractions per day on Days -2 to -1
Drug: Post-transplant Cyclophosphamide (PTCy) — Patients will receive post-transplant cyclophosphamide (PTCy) administered at the dose of 40 mg/kg intravenously on Days +3 to +4.
  Other Names: Cytoxan
Drug: Tacrolimus — Patients will receive tacrolimus administered at a dose adjusted to maintain trough levels between 5-15 ng/mL orally starting on Days +5.
  Other Names: Prograf
Drug: Mycophenolate mofetil (MMF) — Patients will receive mycophenolate mofetil (MMF) administered at the standard dose of 15 mg/kg orally three times daily starting on Day +5 to Day +35 or per institutional guidelines.
  Other Names: CellCept

SUMMARY:
The Flu-TBI 800 trial is a prospective, single-arm, multicenter, interventional phase 2 study to evaluate whether fludarabine plus intermediate-dose total body irradiation (TBI 800 cGy) with post-transplant cyclophosphamide (PTCy) (experimental regimen) improves the 1-year survival of allogeneic stem cell transplant recipients.

DETAILED DESCRIPTION:
Patients who meet all the inclusion criteria for the study will be enrolled to receive a conditioning regimen consisting of fludarabine, administered at a dose of 30 mg/m2 daily on Days -6 to -2, plus intermediate-dose total body irradiation (TBI), administered at a dose of 800 cGy in 4 total fractions, 2 fractions on Days -2 and and 2 fractions on day -1, followed by an infusion of hematopoietic stem cells on Day 0. GVHD prophylaxis will consist of post-transplant cyclophosphamide (PTCy), administered at a dose of 40 mg/kg on Days +3 and +4, as well as tacrolimus (starting on Day +5) and mycophenolate mofetil (on Days +5 to +35).

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 18-65 years.
* Patients with a diagnosis of one of the following hematologic malignancies:
* Acute myeloid leukemia or chronic myeloid leukemia with no circulating blasts and less than 5% blasts in the bone marrow;
* Myelodysplastic syndrome with less than 5% blasts in the bone marrow by IHC or flow cytometry whichever is highest;
* Myeloproliferative neoplasms with less than 5% blast in the marrow and peripheral blood;
* Acute lymphoblastic leukemia in CR (CIBMTR criteria); or Lymphoma in CR (CIBMTR criteria).
* Patients who are eligible for allogeneic stem cell transplant per Transplant Program SOPs.
* Patients with a Karnofsky performance status (KPS) of ≥60%.
* Patients with adequate organ function defined by:

  * Cardiac: LVEF ≥50%
  * Pulmonary: DLCO ≥50% of predicted
  * Hepatic: Bilirubin ≤1.5x ULN, ALT/AST ≤2.5x ULN
  * Renal: Creatinine clearance ≥50 mL/min
* All participants of reproductive potential must use effective contraception following allogeneic hematopoietic stem cell transplantation (allo-HSCT), in accordance with guidelines from the American Society for Transplantation and Cellular Therapy (ASTCT), the FDA, and other expert bodies.
* For Male Participants:

  ○ Male participants must use effective contraception for at least 12 months after transplant, and longer if receiving immunosuppressive or cytotoxic medications. Chemotherapy and radiation can cause DNA damage to sperm, and even if fertility returns, mutations may persist for months. In cases where drugs such as mycophenolate mofetil (MMF) or lenalidomide are used, FDA guidance requires contraception for at least 90 days after discontinuation. Sperm cryopreservation should be offered prior to conditioning. Participants must avoid fathering a child during this time frame.15-17
* For Female Participants:

  * Female participants of childbearing potential are required to use highly effective contraception for a minimum of 12 to 24 months post-transplant, or longer if still receiving immunosuppressive or teratogenic therapy. For drugs such as MMF, sirolimus, or ruxolitinib, contraception must continue for 3 months after the last dose.
  * A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.15-17
* Patients with a suitable donor for allogeneic stem cell transplant defined by:

  * Matched sibling donors willing to donate mobilized peripheral blood (PBSC) or bone marrow (BM), meeting all institutional criteria for donation;
  * Unrelated donors at >7/8 (i.e., mismatched at only one of the HLA-A, HLA-B, HLA-C, and HLA-DRB1 loci) willing to donate mobilized PBSC or BM, and medically eligible to donate cells according to National Marrow Donor Program criteria; or Related Haploidentical donors willing to donate PBSC or BM and meeting criteria for donation.
* Patients who are able to comply with follow-up visits and treatment plans.
* Patients who are able to give informed consent.

Exclusion Criteria:

* Hematopoietic cell transplantation comorbidity index above 3.
* Patients with a Karnofsky performance status (KPS) of <60%.
* Patients with active infections or other contraindications for allogeneic stem cell transplant.
* Patients who are unable or unwilling to give informed consent.
* Patients who have received a prior allogeneic transplant.
* Patients who are unable to comply with follow-up visits and treatment plans.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2032-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) at 1-year following treatment with fludarabine plus intermediate-dose total body irradiation (TBI 800 cGy) with post-transplant cyclophosphamide (PTCy) | Patient status (dead or alive) will be reviewed (e.g., through patient chart review,patient phone call, etc.) up through a period of 1 year
  OS is defined as the time from the first dose of study treatment to the time of death due to any cause. Patients who are still alive will be censored at the date last known alive of the data cut-off date (if applicable), whichever is earlier.

SECONDARY OUTCOMES:
Transplant-related mortality (TRM) at 1-year following treatment with fludarabine plus intermediate-dose total body irradiation (TBI 800 cGy) with post-transplant cyclophosphamide (PTCy) | Patient status (dead or alive) will be reviewed (e.g., through patient chart review,patient phone call, etc.) up through a period of 1 year
  TRM is defined as death due to causes unrelated to the underlying disease. Patients relapsing are censored as surviving at the time of relapse.
Incidence of grade III-IV acute GVHD following treatment with fludarabine plus intermediate-dose total body irradiation (TBI 800 cGy) with post-transplant cyclophosphamide (PTCy) | Patients will be assessed for acute GVHD symptoms weekly from day +7 until day +100. If acute GVHD symptoms remain active after day +100, weekly GVHD documentation will be encouraged until symptom(s) resolution, up through a period of 1 year
  Acute GVHD will be assessed using the Przepiorka criteria,13 Modified Glucksberg/Keystone criteria, and Center for International Blood and Marrow Transplant Research (CIBMTR) severity index (A-D) according to HMH's standard operating procedure (SOP), "Management of Acute Graft versus Host Disease, BMT 500 15."
Incidence of chronic GVHD at 1-year following treatment with fludarabine plus intermediate-dose total body irradiation (TBI 800 cGy) with post-transplant cyclophosphamide (PTCy) | Patients will be assessed for chronic GVHD signs and/or symptoms at a minimum of every three months for the first year post-transplant.
  Chronic GVHD will be assessed based on the 2014 National Institutes of Health (NIH) Consensus Conference Criteria according to HMH's SOP, "Chronic Graft Versus Host Disease, BMT 500 11."
GVHD-free, relapse-free survival (GRFS) at 1-year following treatment with fludarabine plus intermediate-dose total body irradiation (TBI 800 cGy) with post-transplant cyclophosphamide (PTCy) | Patient status (GVHD-free, relapse-free or not) will be reviewed (e.g., throughpatient chart review, patient phone call, etc.) up through a period of 1 year
  GVHD-free, relapse-free survival (GRFS) is a composite endpoint that includes grades 3-4 acute GVHD, chronic GVHD requiring systemic therapy, relapse, or death in the first post-transplant year.
Disease status assessment 2-4 months following treatment with fludarabine plus intermediate-dose total body irradiation (TBI 800 cGy) with post-transplant cyclophosphamide (PTCy) | Patient disease status assessments (e.g., PET-CT, bone marrow, peripheral blood,etc.) will be reviewed (e.g., through patient chart review, etc.) up through a period of 2-4 months following treatment
  Disease status assessment is based on the CIBMTR criterion (see section 8 for more information).
Relapse rate at 1-year following treatment with fludarabine plus intermediate-dose total body irradiation (TBI 800 cGy) with post-transplant cyclophosphamide (PTCy) | Patient status (relapse or continued response) will be reviewed (e.g., throughpatient chart review, patient phone call, etc.) up through a period of 1 year
  Relapse is based on the CIBMTR criterion (see section 8 for more information).
Incidence of Treatment-Emergent Adverse Events with fludarabine plus intermediate-dose total body irradiation (TBI 800 cGy) with post-transplant cyclophosphamide (PTCy) | Following treatment and allogeneic stem cell transplant, all participants will befollowed for safety throughout treatment and the hospital admission as well as longer termsafety follow-up assessments every 3 months for a period of approximately 1 year.
  Adverse events (AEs) will be assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 or severity grade when CTCAE grading does not exist. Grade 1 to 5 will be used to characterize the severity of the AE. If CTCAE grading does not exist for an AE, the severity of mild, moderate, severe, life-threatening and death due to the AE, corresponding respectively to Grades 1 - 5, will be used. This grading system applies except for hematological toxicity where grade 4 cytopenias are anticipated in transplant recipients.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Donato, MD, Principal Investigator — Hackensack Meridian Health
Locations (3):
- United States (3):
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Jersey Shore University Medical Center, Neptune City, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martens MJ, Lian Q, Geller NL, Leifer ES, Logan BR. Sequential monitoring of time-to-event safety endpoints in clinical trials. Clin Trials. 2025 Jun;22(3):267-278. doi: 10.1177/17407745241304119. Epub 2024 Dec 29. PMID 40396502
- [Background] Wu J, Chen L, Wei J, Weiss H, Chauhan A. Two-stage phase II survival trial design. Pharm Stat. 2020 May;19(3):214-229. doi: 10.1002/pst.1983. Epub 2019 Nov 21. PMID 31749311
- [Background] Mycophenolate REMS (Risk Evaluation and Mitigation Strategy). https://www.accessdata.fda.gov
- [Background] Vaxman I, Muchtar E, Jacob E, Kapoor P, Kumar S, Dispenzieri A, Buadi F, Dingli D, Gonsalves W, Kourelis T, Warsame R, Lacy M, Hogan W, Gertz MA. The Efficacy and Safety of Chemotherapy-Based Stem Cell Mobilization in Multiple Myeloma Patients Who Are Poor Responders to Induction: The Mayo Clinic Experience. Transplant Cell Ther. 2021 Sep;27(9):770.e1-770.e7. doi: 10.1016/j.jtct.2021.06.016. Epub 2021 Jun 18. PMID 34153504
- [Background] Xhaard A, Rocha V, Bueno B, de Latour RP, Lenglet J, Petropoulou A, Rodriguez-Otero P, Ribaud P, Porcher R, Socie G, Robin M. Steroid-refractory acute GVHD: lack of long-term improved survival using new generation anticytokine treatment. Biol Blood Marrow Transplant. 2012 Mar;18(3):406-13. doi: 10.1016/j.bbmt.2011.06.012. Epub 2011 Jul 4. PMID 21736868
- [Background] Sengsayadeth S, Wang T, Lee SJ, Haagenson MD, Spellman S, Fernandez Vina MA, Muller CR, Verneris MR, Savani BN, Jagasia M. Cytotoxic T-lymphocyte antigen-4 single nucleotide polymorphisms are not associated with outcomes after unrelated donor transplantation: a center for international blood and marrow transplant research analysis. Biol Blood Marrow Transplant. 2014 Jun;20(6):900-3. doi: 10.1016/j.bbmt.2014.03.005. Epub 2014 Mar 14. PMID 24631737
- [Background] Przepiorka D, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995 Jun;15(6):825-8. PMID 7581076
- [Background] Lee JW, Cho BS, Lee SE, Eom KS, Kim YJ, Kim HJ, Lee S, Min CK, Cho SG, Min WS, Park CW. The Outcome of Unrelated Hematopoietic Stem Cell Transplants with Total Body Irradiation (800 cGy) and Cyclophosphamide (120 mg/kg) in Adult Patients with Acquired Severe Aplastic Anemia. Biol Blood Marrow Transplant. 2011 Jan;17(1):101-8. doi: 10.1016/j.bbmt.2010.06.014. Epub 2010 Jun 25. PMID 20601037
- [Background] Sanchez-Petitto G, Huang Y, Bezerra E, et al. Comparison of Two Myeloablative Total-Body Irradiation (MAC-TBI) Regimens: 1200 Cgy Vs 800 Cgy of TBI for Allogeneic Stem Cell Transplantation in Adults with Hematological Malignancies. Blood. 2024;144(Supplement 1):7303-7303. doi:10.1182/blood-2024-194146
- [Background] Sterling CH, Hughes MS, Tsai HL, et al. Non-myeloablative allogeneic blood or marrow transplantation (AlloBMT) with post-transplant cyclophosphamide (PTCy) for peripheral T- cell lymphoma (PTCL): Improved outcomes with peripheral blood (PB) allografts and increased total body irradiation (TBI) to 400 cGV. J Clin Oncol. 2022;40(16_suppl):7047- 7047. doi:10.1200/JCO.2022.40.16_suppl.7047
- [Background] Gooley TA, Chien JW, Pergam SA, Hingorani S, Sorror ML, Boeckh M, Martin PJ, Sandmaier BM, Marr KA, Appelbaum FR, Storb R, McDonald GB. Reduced mortality after allogeneic hematopoietic-cell transplantation. N Engl J Med. 2010 Nov 25;363(22):2091-101. doi: 10.1056/NEJMoa1004383. PMID 21105791
- [Background] Ciurea S, Zhang M, Kanakry C. CNIs versus post-transplant cyclophosphamide-based GVHD prophylaxis in haploidentical transplantation. Blood. 2020;137(4):444-455.
- [Background] Kanakry CG, Tsai HL, Bolanos-Meade J, Smith BD, Gojo I, Kanakry JA, Kasamon YL, Gladstone DE, Matsui W, Borrello I, Huff CA, Swinnen LJ, Powell JD, Pratz KW, DeZern AE, Showel MM, McDevitt MA, Brodsky RA, Levis MJ, Ambinder RF, Fuchs EJ, Rosner GL, Jones RJ, Luznik L. Single-agent GVHD prophylaxis with posttransplantation cyclophosphamide after myeloablative, HLA-matched BMT for AML, ALL, and MDS. Blood. 2014 Dec 11;124(25):3817-27. doi: 10.1182/blood-2014-07-587477. Epub 2014 Oct 14. PMID 25316679
- [Background] Bolanos-Meade J, Hamadani M, Wu J, Al Malki MM, Martens MJ, Runaas L, Elmariah H, Rezvani AR, Gooptu M, Larkin KT, Shaffer BC, El Jurdi N, Loren AW, Solh M, Hall AC, Alousi AM, Jamy OH, Perales MA, Yao JM, Applegate K, Bhatt AS, Kean LS, Efebera YA, Reshef R, Clark W, DiFronzo NL, Leifer E, Horowitz MM, Jones RJ, Holtan SG; BMT CTN 1703 Investigators. Post-Transplantation Cyclophosphamide-Based Graft-versus-Host Disease Prophylaxis. N Engl J Med. 2023 Jun 22;388(25):2338-2348. doi: 10.1056/NEJMoa2215943. PMID 37342922
- [Background] Luznik L, O'Donnell PV, Fuchs EJ. Post-transplantation cyclophosphamide for tolerance induction in HLA-haploidentical bone marrow transplantation. Semin Oncol. 2012 Dec;39(6):683-93. doi: 10.1053/j.seminoncol.2012.09.005. PMID 23206845
- [Background] Scott BL, Pasquini MC, Logan BR, Wu J, Devine SM, Porter DL, Maziarz RT, Warlick ED, Fernandez HF, Alyea EP, Hamadani M, Bashey A, Giralt S, Geller NL, Leifer E, Le-Rademacher J, Mendizabal AM, Horowitz MM, Deeg HJ, Horwitz ME. Myeloablative Versus Reduced-Intensity Hematopoietic Cell Transplantation for Acute Myeloid Leukemia and Myelodysplastic Syndromes. J Clin Oncol. 2017 Apr 10;35(11):1154-1161. doi: 10.1200/JCO.2016.70.7091. Epub 2017 Feb 13. PMID 28380315
- [Background] Copelan EA. Hematopoietic stem-cell transplantation. N Engl J Med. 2006 Apr 27;354(17):1813-26. doi: 10.1056/NEJMra052638. No abstract available. PMID 16641398
- [Background] Baron F, Labopin M, Blaise D. Reduced-intensity conditioning versus myeloablative conditioning allogeneic hematopoietic stem cell transplantation in acute myeloid leukemia: A study from the Acute Leukemia Working Party of the EBMT. Blood. 2017;129(4):448-456.
- [Background] Gyurkocza B, Rezvani A, Storb RF. Allogeneic hematopoietic cell transplantation: the state of the art. Expert Rev Hematol. 2010 Jun;3(3):285-99. doi: 10.1586/ehm.10.21. PMID 20871781